CLINICAL TRIAL: NCT06864260
Title: Cancer PRevention Through Enhanced EnvironMenT
Acronym: PREEMpT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lori Bateman, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300011733; 5U54CA280770-02 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cancer Risk
Keywords: cancer; persistent poverty; built environment; social determinants of health; social environment; allostatic load; collective efficacy; perceived stress; cancer screening; neighborhood safety
MeSH Terms: conditions — Neoplasms | interventions — Built Environment

STUDY DESIGN:
Intervention Model Description: Using a sequential explanatory mixed methods design, quantitative (surveys) and qualitative (focus groups) data will be collected to assess community-level changes in perceptions and behaviors in targeted census tracts. To measure chronic stress objectively (as a proxy for cancer risk), study staff will draw blood to measure stress biomarkers, which will include 10 indicators of allostatic load. A two-group design with independent, mutually exclusive samples pre- and post-intervention will be utilized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-Intervention Group (No Intervention): Baseline data will be collected on participants in this arm before community-level built and social environment modifications (intervention) are implemented.
- Post-Intervention Group (Experimental): Post-intervention data will be collected on participants in this arm (different participants than in the pre-intervention group) after community-level built and social environment modifications (intervention) are implemented.
  Interventions: Other: Built Environment; Other: Social Environment

INTERVENTIONS:
Other: Built Environment — Built environment modifications include sidewalks, sidewalk cuts, traffic-calming devices, crosswalks, transit improvements, green space, street trees, beautification, signage, lighting, wellness van
  Arms: Post-Intervention Group
Other: Social Environment — Neighborhood coalition, Community Leadership Academy (LHSA), community-led events, community health workers
  Arms: Post-Intervention Group

SUMMARY:
The goal of Cancer PRevention through Enhanced EnvironMenT (Cancer PREEMpT) is to test whether a comprehensive intervention that improves the neighborhood built and social environment can reduce community-level cancer risk in persistent poverty (PP) areas. Our overall hypothesis is that enhancements of the living environment (both built and social) will lower cancer risk through several mechanisms. Built environment improvements will impact walkability (through improved lighting, sidewalks, green space) and access to preventive care (through a mobile wellness van and community health workers), which will stimulate health-related behaviors (physical activity, cancer screening). These improvements will also positively impact safety (through blight removal, traffic calming), social cohesion (through opportunities for socialization), and collective efficacy (through improved neighborhood perceptions). Social environment improvements will increase social cohesion (through community-led events) and collective efficacy (through a Community Leadership Academy and community grants), which will improve public safety as well as facilitate health-related behaviors (physical activity, prevention/wellness). Both types of improvements (built and social environment) will help reduce chronic stress, which will lower the PP community's cancer risk.

DETAILED DESCRIPTION:
Disparities in cancer prevention and outcomes by poverty status are well documented. Such disparities are rooted in structural and intermediate social determinants of health (SDOH), including neighborhood built and social environment (together referred to as living environment). Features of the living environment have major implications for cancer risk through behaviors such as physical activity and access to preventive care. Adverse neighborhood conditions also exacerbate the stress response, in the form of high allostatic load, which is a risk factor for many cancers. Reducing cancer disparities in persistent poverty (PP) areas requires a multisectoral approach in which citizens, organizations, businesses, and local governments unite to improve neighborhood conditions. However, despite compelling evidence that the living environment impacts health-related behaviors and outcomes, including cancer, there are virtually no interventions that determine to what extent modifications of the neighborhood built and social environments reduce cancer risk. Based on the Alcarez framework, the proposed study aims to fill this knowledge gap. The purpose of the study is to understand if interventions aimed at improving neighborhood built and social environment can reduce community-level cancer risk in 5 targeted PP neighborhoods (census tracts). Study specific aims are as follows:

Aim 1. Implement Cancer PREEMpT and assess whether the enhancement of living environment leads to increased public safety, use of parks and community spaces, community events, and prevention services.

After a community-engaged needs assessment, built and social environment improvements will be implemented in collaboration with our study partner, Live HealthSmart Alabama (LHSA). Public usage data will be gathered regarding public safety, use of parks and community spaces, and community events. The LHSA wellness van will visit PREEMpT targeted communities on a monthly basis for preventive assessments and referrals to primary care and cancer screening (cervical, breast, and colon). The public usage data will be gathered through non-human subjects (numeric counts, public crime data, and civil data). The prevention data will be gathered by the LHSA wellness van staff through de-identified counts of uptake of services by community members.

Aim 2. Determine the effect of improved living environment on community-level perceptions and behaviors related to cancer risk.

Using a sequential explanatory mixed methods design, surveys will be collected and focus groups will be conducted to assess community-level changes in perceptions and behaviors in the targeted areas. For the quantitative (survey) component, a two-group survey design will be used with independent, mutually exclusive samples pre- and post-intervention, and for the qualitative (focus group) component, focus groups with residents pre- and post-intervention will be conducted.

(2.1) SURVEYS. Surveys will be conducted with 150 participants from the targeted areas at baseline and 150 surveys with another set of participants from the targeted area in the last year of the study. The surveys will be administered by the staff of UAB Recruitment and Retention Shared Facility (RRSF).

(2.2) FOCUS GROUPS: 3 focus groups will be conducted at baseline and in the last year of the project, with approximately 6-10 participants per group. Participants will be randomly selected from those who complete pre- and post-intervention surveys (in 2.1 above). Focus groups will be moderated by trained staff who will a use semi-structured focus group guide to explore external barriers, facilitators, and community cultural norms associated with physical activity, safety, and wellness, with an emphasis on cancer prevention. Participants will also discuss factors related to the neighborhood built environment, social environment, and perceptions of crime.

Aim 3. Evaluate the impact of improved living environments on perceived and objective chronic stress.

Perceived Stress - Self-reported stress will be measured with the Perceived Stress Scale included in the Aim 2 surveys.

Objective Chronic Stress - Blood will be drawn in a sub-sample of participants to measure stress biomarkers, which will include 10 measures of allostatic load (AL). To assess community-level changes in AL, an experimental two-group design will be used with independent, mutually exclusive samples at baseline and Year 5. At baseline, 50 participants from the 150 survey respondents enrolled in the pre-intervention group (Aim 2) will be randomly selected, and at Year 5, 50 participants from the 150 survey respondents enrolled in the post-intervention group (Aim 2) will be randomly selected (for a total N = 100).

ELIGIBILITY:
Inclusion Criteria:

* Black race
* English speaker
* Resident of targeted census tract

Exclusion Criteria:

* Non Black race
* Non-English speaker
* Not a resident of targeted community

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with High Allostatic Load | baseline, up to 3 years
  10 indicators that make up allostatic load (AL) score, a measure of the cumulative burden of stress. The AL score is defined as sum score of the number of biomarkers that are above the set threshold, with a high level being 3 or more biomarkers above the threshold.
Average Level of Perceived Stress Among Participants | baseline, up to 3 years
  10-item Perceived Stress Scale (PSS) which asks about the person's feelings and thoughts during the past month and their frequency (0=Never; 1=Almost Never; 2=Sometimes; 3=Fairly Often; 4=Very Often)

SECONDARY OUTCOMES:
Average Self-Reported Leisure Time Physical Activity Among Participants | baseline, up to 3 years
  The International Physical Activity Questionnaire (IPAQ) is a 7-item questionnaire of a subject's physical activity over the last 7 days and assesses the types of intensity of physical activity and sitting time that people do as part of daily living. Estimates the total physical activity in MET-min/week and time spent sitting.
Average Healthy Food Access among Participants | baseline, up to 3 years
  The Perceived Availability of Healthy Foods Scale is estimated by taking the average across the three items. Lower mean scores indicate better availability of healthy foods (i.e., low-fat products, fruits, and vegetables) within a 20 minute walk from home.
Cancer screening frequency among participants | baseline, up to 3 years
  Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial, Baseline Questionnaire for Male (BQMC) & Female (BQM3) includes 10 questions (8 for women and 5 for men) that ask about cancer screening tests that a respondent has had in the past 3 years.
Average Social Support among Participants | baseline, up to 3 years
  Social support from Medical Outcomes Study (RAND) consists of 19 questions with Likert scale responses. The survey consists of an overall functional social support index. A higher score indicates more support. To obtain an overall support index, the average of the scores for all19 items included is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lori B Bateman, PhD, Principal Investigator — University of Alabama at Birmingham; Gabriela R Oates, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication, after de-identification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 3 months to 5 years after publication date
Access Criteria: Deidentified individual data that supports publication results will be shared beginning 3 months and up to 60 months following publication, provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UAB.

REFERENCES:
- [Background] Rodriquez EJ, Kim EN, Sumner AE, Napoles AM, Perez-Stable EJ. Allostatic Load: Importance, Markers, and Score Determination in Minority and Disparity Populations. J Urban Health. 2019 Mar;96(Suppl 1):3-11. doi: 10.1007/s11524-019-00345-5. PMID 30671711
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cerin E, Saelens BE, Sallis JF, Frank LD. Neighborhood Environment Walkability Scale: validity and development of a short form. Med Sci Sports Exerc. 2006 Sep;38(9):1682-91. doi: 10.1249/01.mss.0000227639.83607.4d. PMID 16960531
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Pearlin LI, Bierman A. Current Issues and Future Directions in Research into the Stress Process. In: C.S. A, J.C. P, A. B, eds. Handbook of the Sociology of Mental Health. Springer; 2013:325-340.
- [Background] Alcaraz KI, Wiedt TL, Daniels EC, Yabroff KR, Guerra CE, Wender RC. Understanding and addressing social determinants to advance cancer health equity in the United States: A blueprint for practice, research, and policy. CA Cancer J Clin. 2020 Jan;70(1):31-46. doi: 10.3322/caac.21586. Epub 2019 Oct 29. PMID 31661164
- [Background] Gomez SL, Shariff-Marco S, DeRouen M, Keegan TH, Yen IH, Mujahid M, Satariano WA, Glaser SL. The impact of neighborhood social and built environment factors across the cancer continuum: Current research, methodological considerations, and future directions. Cancer. 2015 Jul 15;121(14):2314-30. doi: 10.1002/cncr.29345. Epub 2015 Apr 6. PMID 25847484
- [Background] Shariff-Marco S, Von Behren J, Reynolds P, Keegan TH, Hertz A, Kwan ML, Roh JM, Thomsen C, Kroenke CH, Ambrosone C, Kushi LH, Gomez SL. Impact of Social and Built Environment Factors on Body Size among Breast Cancer Survivors: The Pathways Study. Cancer Epidemiol Biomarkers Prev. 2017 Apr;26(4):505-515. doi: 10.1158/1055-9965.EPI-16-0932. Epub 2017 Feb 2. PMID 28154107
- [Background] Lynch SM, Handorf E, Sorice KA, Blackman E, Bealin L, Giri VN, Obeid E, Ragin C, Daly M. The effect of neighborhood social environment on prostate cancer development in black and white men at high risk for prostate cancer. PLoS One. 2020 Aug 13;15(8):e0237332. doi: 10.1371/journal.pone.0237332. eCollection 2020. PMID 32790761
- [Background] Frank LD, Saelens BE, Powell KE, Chapman JE. Stepping towards causation: do built environments or neighborhood and travel preferences explain physical activity, driving, and obesity? Soc Sci Med. 2007 Nov;65(9):1898-914. doi: 10.1016/j.socscimed.2007.05.053. Epub 2007 Jul 17. PMID 17644231
- [Background] Obeng-Gyasi S, Tarver W, Carlos RC, Andersen BL. Allostatic load: a framework to understand breast cancer outcomes in Black women. NPJ Breast Cancer. 2021 Jul 30;7(1):100. doi: 10.1038/s41523-021-00309-6. No abstract available. PMID 34330927
- [Background] Akinyemiju T, Wilson LE, Deveaux A, Aslibekyan S, Cushman M, Gilchrist S, Safford M, Judd S, Howard V. Association of Allostatic Load with All-Cause andCancer Mortality by Race and Body Mass Index in theREGARDS Cohort. Cancers (Basel). 2020 Jun 26;12(6):1695. doi: 10.3390/cancers12061695. PMID 32604717
- [Background] McEwen BS, Stellar E. Stress and the individual. Mechanisms leading to disease. Arch Intern Med. 1993 Sep 27;153(18):2093-101. PMID 8379800